CLINICAL TRIAL: NCT04540926
Title: Utility of Low Doses of Corticosteroids and Cyclosporine Combined With Enoxaparin, in Patients With COVID-19 Pneumonia at the ISSSTE Regional Hospital, Puebla, During the Contingency Period Due to the SARS-Cov2 Pandemic
Brief Title: Cyclosporine A Plus Low-steroid Treatment in COVID-19 Pneumonia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado (Other Government)
Responsible Party: Principal Investigator, JOSE LUIS GALVEZ-ROMERO, Master in Medical Sciences and Reasearch and Medical Doctor, Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 135.2020
Record Dates: First submitted 2020-09-02; First posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: COVID 19 Pneumonia
MeSH Terms: interventions — Cyclosporine

STUDY DESIGN:
Intervention Model Description: Consecutive patients with suspected or confirmed diagnosis of COVID-19 were assigned, in an unblinded and non-randomized fashion, to receive either steroids plus CsA (intervention group) or steroids only (standard of treatment in this hospital, control group), as per individual clinical judgment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COVID-19 Pneumonia control group (Experimental): COVID-19 pneumonia patients with standar treatment: enoxaparin 0.5 mg/kg S.C. once, Clarithromycin 500 mg twice an metylprednisolone 0.5 mg/kg once endovenous.
  Interventions: Drug: Cyclosporin A

INTERVENTIONS:
Drug: Cyclosporin A — COVID-19 pneumonia patients treated with oral CsA at a dose of 1-2 mg /kg / day divided into two doses, for 7 days, since entering to hospitalization.

SUMMARY:
Methods: Single-center pilot study included PCR+ SARS-CoV2-patients, hospitalized from April to May 2020 in Puebla, Mexico. Comparative treatment with steroids plus CsA or steroids. Mild, moderate or severe pneumonia was measured by clinical, laboratory tests, lung damage score by computed tomography, and score for clinical improvement. Death rate was evaluated at 28 days.

DETAILED DESCRIPTION:
This is a pilot study done in a single center (ISSSTE Regional Hospital, Puebla, Mexico). Consecutive patients with suspected or confirmed diagnosis of COVID-19 were assigned, in an unblinded and non-randomized fashion, to receive either steroids plus CsA (intervention group) or steroids only (standard of treatment in this hospital, control group), as per individual clinical judgment. The primary outcome was the number of days to clinical improvement until hospital discharge or death. The secondary outcome was the improvement of patients, defined by the following parameters: lower oxygen requirements (2 liters per minute, or less), absence of fever by three consecutive days, respiratory rate <22, a decrease of 50% or more in the C reactive protein on admission, and length of hospital stay.

Adult patients attending to the hospital between April 15, to May 31, 2020, fulfilling symptoms compatible with COVID-19 pneumonia, according to the WHO guidance, were invited to participate and all the patients gave their written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COVID 19 pneumonia by clinical, lung computed Tomography and RT-PCR nasopharyngeal swabs.

Exclusion Criteria:

* Influenza infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of days to clinical improvement until hospital discharge or death. | 28 days.
  Improvement of patients, defined by the following parameters: lower oxygen requirements (2 liters per minute, or less), absence of fever by three consecutive days, respiratory rate <22, a decrease of 50% or more in the C reactive protein on admission, and length of hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: JOSE LUIS J GALVEZ-ROMERO, MD, Principal Investigator — Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado
Locations (1):
- Jose Luis Jl Galvez-Romero, Puebla City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fehr AR, Perlman S. Coronaviruses: an overview of their replication and pathogenesis. Methods Mol Biol. 2015;1282:1-23. doi: 10.1007/978-1-4939-2438-7_1. PMID 25720466
- [Result] Lake MA. What we know so far: COVID-19 current clinical knowledge and research. Clin Med (Lond). 2020 Mar;20(2):124-127. doi: 10.7861/clinmed.2019-coron. Epub 2020 Mar 5. PMID 32139372
- [Result] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Result] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Result] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Result] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Result] Jamilloux Y, Henry T, Belot A, Viel S, Fauter M, El Jammal T, Walzer T, Francois B, Seve P. Should we stimulate or suppress immune responses in COVID-19? Cytokine and anti-cytokine interventions. Autoimmun Rev. 2020 Jul;19(7):102567. doi: 10.1016/j.autrev.2020.102567. Epub 2020 May 4. PMID 32376392
- [Result] Kupferschmidt K, Cohen J. Race to find COVID-19 treatments accelerates. Science. 2020 Mar 27;367(6485):1412-1413. doi: 10.1126/science.367.6485.1412. No abstract available. PMID 32217705
- [Result] Russell CD, Millar JE, Baillie JK. Clinical evidence does not support corticosteroid treatment for 2019-nCoV lung injury. Lancet. 2020 Feb 15;395(10223):473-475. doi: 10.1016/S0140-6736(20)30317-2. Epub 2020 Feb 7. No abstract available. PMID 32043983
- [Result] Villar J, Belda J, Anon JM, Blanco J, Perez-Mendez L, Ferrando C, Martinez D, Soler JA, Ambros A, Munoz T, Rivas R, Corpas R, Diaz-Dominguez FJ, Soro M, Garcia-Bello MA, Fernandez RL, Kacmarek RM; DEXA-ARDS Network. Evaluating the efficacy of dexamethasone in the treatment of patients with persistent acute respiratory distress syndrome: study protocol for a randomized controlled trial. Trials. 2016 Jul 22;17:342. doi: 10.1186/s13063-016-1456-4. PMID 27449641
- [Result] Lamontagne F, Rochwerg B, Lytvyn L, Guyatt GH, Moller MH, Annane D, Kho ME, Adhikari NKJ, Machado F, Vandvik PO, Dodek P, Leboeuf R, Briel M, Hashmi M, Camsooksai J, Shankar-Hari M, Baraki MK, Fugate K, Chua S, Marti C, Cohen D, Botton E, Agoritsas T, Siemieniuk RAC. Corticosteroid therapy for sepsis: a clinical practice guideline. BMJ. 2018 Aug 10;362:k3284. doi: 10.1136/bmj.k3284. No abstract available. PMID 30097460
- [Result] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Result] Shang L, Zhao J, Hu Y, Du R, Cao B. On the use of corticosteroids for 2019-nCoV pneumonia. Lancet. 2020 Feb 29;395(10225):683-684. doi: 10.1016/S0140-6736(20)30361-5. Epub 2020 Feb 12. No abstract available. PMID 32122468
- [Result] RECOVERY Collaborative Group; Horby P, Lim WS, Emberson JR, Mafham M, Bell JL, Linsell L, Staplin N, Brightling C, Ustianowski A, Elmahi E, Prudon B, Green C, Felton T, Chadwick D, Rege K, Fegan C, Chappell LC, Faust SN, Jaki T, Jeffery K, Montgomery A, Rowan K, Juszczak E, Baillie JK, Haynes R, Landray MJ. Dexamethasone in Hospitalized Patients with Covid-19. N Engl J Med. 2021 Feb 25;384(8):693-704. doi: 10.1056/NEJMoa2021436. Epub 2020 Jul 17. PMID 32678530
- [Result] Zeidler HK, Kvien TK, Hannonen P, Wollheim FA, Forre O, Geidel H, Hafstrom I, Kaltwasser JP, Leirisalo-Repo M, Manger B, Laasonen L, Markert ER, Prestele H, Kurki P. Progression of joint damage in early active severe rheumatoid arthritis during 18 months of treatment: comparison of low-dose cyclosporin and parenteral gold. Br J Rheumatol. 1998 Aug;37(8):874-82. doi: 10.1093/rheumatology/37.8.874. PMID 9734679
- [Result] Tokuda M, Kurata N, Mizoguchi A, Inoh M, Seto K, Kinashi M, Takahara J. Effect of low-dose cyclosporin A on systemic lupus erythematosus disease activity. Arthritis Rheum. 1994 Apr;37(4):551-8. doi: 10.1002/art.1780370416. PMID 8147933
- [Result] Liddicoat AM, Lavelle EC. Modulation of innate immunity by cyclosporine A. Biochem Pharmacol. 2019 May;163:472-480. doi: 10.1016/j.bcp.2019.03.022. Epub 2019 Mar 15. PMID 30880061
- [Result] Li HS, Kuok DIT, Cheung MC, Ng MMT, Ng KC, Hui KPY, Peiris JSM, Chan MCW, Nicholls JM. Effect of interferon alpha and cyclosporine treatment separately and in combination on Middle East Respiratory Syndrome Coronavirus (MERS-CoV) replication in a human in-vitro and ex-vivo culture model. Antiviral Res. 2018 Jul;155:89-96. doi: 10.1016/j.antiviral.2018.05.007. Epub 2018 May 17. PMID 29772254
- [Result] Tanaka Y, Sato Y, Sasaki T. Suppression of coronavirus replication by cyclophilin inhibitors. Viruses. 2013 May 22;5(5):1250-60. doi: 10.3390/v5051250. PMID 23698397
- [Result] de Wilde AH, Zevenhoven-Dobbe JC, van der Meer Y, Thiel V, Narayanan K, Makino S, Snijder EJ, van Hemert MJ. Cyclosporin A inhibits the replication of diverse coronaviruses. J Gen Virol. 2011 Nov;92(Pt 11):2542-2548. doi: 10.1099/vir.0.034983-0. Epub 2011 Jul 13. PMID 21752960
- [Result] Wang Y, Dong C, Hu Y, Li C, Ren Q, Zhang X, Shi H, Zhou M. Temporal Changes of CT Findings in 90 Patients with COVID-19 Pneumonia: A Longitudinal Study. Radiology. 2020 Aug;296(2):E55-E64. doi: 10.1148/radiol.2020200843. Epub 2020 Mar 19. PMID 32191587
- [Result] Ji D, Zhang D, Xu J, Chen Z, Yang T, Zhao P, Chen G, Cheng G, Wang Y, Bi J, Tan L, Lau G, Qin E. Prediction for Progression Risk in Patients With COVID-19 Pneumonia: The CALL Score. Clin Infect Dis. 2020 Sep 12;71(6):1393-1399. doi: 10.1093/cid/ciaa414. PMID 32271369
- [Result] Wiersinga WJ, Rhodes A, Cheng AC, Peacock SJ, Prescott HC. Pathophysiology, Transmission, Diagnosis, and Treatment of Coronavirus Disease 2019 (COVID-19): A Review. JAMA. 2020 Aug 25;324(8):782-793. doi: 10.1001/jama.2020.12839. PMID 32648899
- [Result] Annane D, Renault A, Bellissant E. Glucocorticoids with or without Fludrocortisone in Septic Shock. N Engl J Med. 2018 Aug 30;379(9):895-6. doi: 10.1056/NEJMc1804993. No abstract available. PMID 30179381
- [Result] Venkatesh B, Finfer S, Myburgh J; ADRENAL investigators. Glucocorticoids with or without Fludrocortisone in Septic Shock. N Engl J Med. 2018 Aug 30;379(9):895. doi: 10.1056/NEJMc1804993. No abstract available. PMID 30157400
- [Result] Alhazzani W, Moller MH, Arabi YM, Loeb M, Gong MN, Fan E, Oczkowski S, Levy MM, Derde L, Dzierba A, Du B, Aboodi M, Wunsch H, Cecconi M, Koh Y, Chertow DS, Maitland K, Alshamsi F, Belley-Cote E, Greco M, Laundy M, Morgan JS, Kesecioglu J, McGeer A, Mermel L, Mammen MJ, Alexander PE, Arrington A, Centofanti JE, Citerio G, Baw B, Memish ZA, Hammond N, Hayden FG, Evans L, Rhodes A. Surviving Sepsis Campaign: guidelines on the management of critically ill adults with Coronavirus Disease 2019 (COVID-19). Intensive Care Med. 2020 May;46(5):854-887. doi: 10.1007/s00134-020-06022-5. Epub 2020 Mar 28. PMID 32222812
- [Result] Wong SS, Yuen KY. The management of coronavirus infections with particular reference to SARS. J Antimicrob Chemother. 2008 Sep;62(3):437-41. doi: 10.1093/jac/dkn243. Epub 2008 Jun 18. PMID 18565970
- [Result] Lee N, Allen Chan KC, Hui DS, Ng EK, Wu A, Chiu RW, Wong VW, Chan PK, Wong KT, Wong E, Cockram CS, Tam JS, Sung JJ, Lo YM. Effects of early corticosteroid treatment on plasma SARS-associated Coronavirus RNA concentrations in adult patients. J Clin Virol. 2004 Dec;31(4):304-9. doi: 10.1016/j.jcv.2004.07.006. PMID 15494274
- [Result] Arabi YM, Mandourah Y, Al-Hameed F, Sindi AA, Almekhlafi GA, Hussein MA, Jose J, Pinto R, Al-Omari A, Kharaba A, Almotairi A, Al Khatib K, Alraddadi B, Shalhoub S, Abdulmomen A, Qushmaq I, Mady A, Solaiman O, Al-Aithan AM, Al-Raddadi R, Ragab A, Balkhy HH, Al Harthy A, Deeb AM, Al Mutairi H, Al-Dawood A, Merson L, Hayden FG, Fowler RA; Saudi Critical Care Trial Group. Corticosteroid Therapy for Critically Ill Patients with Middle East Respiratory Syndrome. Am J Respir Crit Care Med. 2018 Mar 15;197(6):757-767. doi: 10.1164/rccm.201706-1172OC. PMID 29161116
- [Result] Russell B, Moss C, George G, Santaolalla A, Cope A, Papa S, Van Hemelrijck M. Associations between immune-suppressive and stimulating drugs and novel COVID-19-a systematic review of current evidence. Ecancermedicalscience. 2020 Mar 27;14:1022. doi: 10.3332/ecancer.2020.1022. eCollection 2020. PMID 32256705
- [Result] Zhao Z, Zhang F, Xu M, Huang K, Zhong W, Cai W, Yin Z, Huang S, Deng Z, Wei M, Xiong J, Hawkey PM. Description and clinical treatment of an early outbreak of severe acute respiratory syndrome (SARS) in Guangzhou, PR China. J Med Microbiol. 2003 Aug;52(Pt 8):715-720. doi: 10.1099/jmm.0.05320-0. PMID 12867568
- [Result] Fadel R, Morrison AR, Vahia A, Smith ZR, Chaudhry Z, Bhargava P, Miller J, Kenney RM, Alangaden G, Ramesh MS; Henry Ford COVID-19 Management Task Force. Early Short-Course Corticosteroids in Hospitalized Patients With COVID-19. Clin Infect Dis. 2020 Nov 19;71(16):2114-2120. doi: 10.1093/cid/ciaa601. PMID 32427279
- [Result] Fernandez-Cruz A, Ruiz-Antoran B, Munez-Rubio E, Sancho-Lopez A, Callejas-Diaz A, Avendano-Sola C, Ramos-Martinez A. The Right Time for Steroids in COVID-19. Clin Infect Dis. 2021 Apr 26;72(8):1486-1487. doi: 10.1093/cid/ciaa865. No abstract available. PMID 32585016
- [Result] Selvaraj V, Dapaah-Afriyie K, Finn A, Flanigan TP. Short-Term Dexamethasone in Sars-CoV-2 Patients. R I Med J (2013). 2020 Jun 19;103(6):39-43. PMID 32570995
- [Result] Cour M, Ovize M, Argaud L. Cyclosporine A: a valid candidate to treat COVID-19 patients with acute respiratory failure? Crit Care. 2020 Jun 2;24(1):276. doi: 10.1186/s13054-020-03014-1. No abstract available. PMID 32487139
- [Result] Argaud L, Cour M, Dubien PY, Giraud F, Jossan C, Riche B, Hernu R, Darmon M, Poncelin Y, Tchenio X, Quenot JP, Freysz M, Kamga C, Beuret P, Usseglio P, Badet M, Anette B, Chaulier K, Alasan E, Sadoune S, Bobbia X, Zeni F, Gueugniaud PY, Robert D, Roy P, Ovize M; CYRUS Study Group. Effect of Cyclosporine in Nonshockable Out-of-Hospital Cardiac Arrest: The CYRUS Randomized Clinical Trial. JAMA Cardiol. 2016 Aug 1;1(5):557-65. doi: 10.1001/jamacardio.2016.1701. PMID 27433815
- [Result] Cung TT, Morel O, Cayla G, Rioufol G, Garcia-Dorado D, Angoulvant D, Bonnefoy-Cudraz E, Guerin P, Elbaz M, Delarche N, Coste P, Vanzetto G, Metge M, Aupetit JF, Jouve B, Motreff P, Tron C, Labeque JN, Steg PG, Cottin Y, Range G, Clerc J, Claeys MJ, Coussement P, Prunier F, Moulin F, Roth O, Belle L, Dubois P, Barragan P, Gilard M, Piot C, Colin P, De Poli F, Morice MC, Ider O, Dubois-Rande JL, Unterseeh T, Le Breton H, Beard T, Blanchard D, Grollier G, Malquarti V, Staat P, Sudre A, Elmer E, Hansson MJ, Bergerot C, Boussaha I, Jossan C, Derumeaux G, Mewton N, Ovize M. Cyclosporine before PCI in Patients with Acute Myocardial Infarction. N Engl J Med. 2015 Sep 10;373(11):1021-31. doi: 10.1056/NEJMoa1505489. Epub 2015 Aug 30. PMID 26321103
- [Result] Kreitmann L, Argaud L, Ovize M, Cour M; CYRUS Study Group. Cyclosporine A prevents cardiac arrest-induced acute respiratory failure: a post-hoc analysis of the CYRUS trial. Intensive Care Med. 2020 Jun;46(6):1281-1283. doi: 10.1007/s00134-020-06043-0. Epub 2020 Apr 21. No abstract available. PMID 32318777
- [Result] Naesens M, Kuypers DR, Sarwal M. Calcineurin inhibitor nephrotoxicity. Clin J Am Soc Nephrol. 2009 Feb;4(2):481-508. doi: 10.2215/CJN.04800908. PMID 19218475
- [Result] Sanchez-Pernaute O, Romero-Bueno FI, Selva-O'Callaghan A. Why choose cyclosporin A as first-line therapy in COVID-19 pneumonia. Reumatol Clin. 2021 Nov;17(9):555-557. doi: 10.1016/j.reuma.2020.03.001. Epub 2020 Apr 16. No abstract available. PMID 32354685
- [Result] Pino-Lagos K, Michea P, Sauma D, Alba A, Morales J, Bono MR, Fierro A, Rosemblatt M. Cyclosporin A-treated dendritic cells may affect the outcome of organ transplantation by decreasing CD4+CD25+ regulatory T cell proliferation. Biol Res. 2010;43(3):333-7. Epub 2010 Nov 30. PMID 21249305
- [Result] Greenblatt MB, Aliprantis A, Hu B, Glimcher LH. Calcineurin regulates innate antifungal immunity in neutrophils. J Exp Med. 2010 May 10;207(5):923-31. doi: 10.1084/jem.20092531. Epub 2010 Apr 26. PMID 20421389
- [Result] Roilides E, Robinson T, Sein T, Pizzo PA, Walsh TJ. In vitro and ex vivo effects of cyclosporin A on phagocytic host defenses against Aspergillus fumigatus. Antimicrob Agents Chemother. 1994 Dec;38(12):2883-8. doi: 10.1128/AAC.38.12.2883. PMID 7695277
- [Result] Gupta AK, Giaglis S, Hasler P, Hahn S. Efficient neutrophil extracellular trap induction requires mobilization of both intracellular and extracellular calcium pools and is modulated by cyclosporine A. PLoS One. 2014 May 12;9(5):e97088. doi: 10.1371/journal.pone.0097088. eCollection 2014. PMID 24819773
- [Result] Edler C, Schroder AS, Aepfelbacher M, Fitzek A, Heinemann A, Heinrich F, Klein A, Langenwalder F, Lutgehetmann M, Meissner K, Puschel K, Schadler J, Steurer S, Mushumba H, Sperhake JP. Dying with SARS-CoV-2 infection-an autopsy study of the first consecutive 80 cases in Hamburg, Germany. Int J Legal Med. 2020 Jul;134(4):1275-1284. doi: 10.1007/s00414-020-02317-w. Epub 2020 Jun 4. PMID 32500199
- [Result] Barnes BJ, Adrover JM, Baxter-Stoltzfus A, Borczuk A, Cools-Lartigue J, Crawford JM, Dassler-Plenker J, Guerci P, Huynh C, Knight JS, Loda M, Looney MR, McAllister F, Rayes R, Renaud S, Rousseau S, Salvatore S, Schwartz RE, Spicer JD, Yost CC, Weber A, Zuo Y, Egeblad M. Targeting potential drivers of COVID-19: Neutrophil extracellular traps. J Exp Med. 2020 Jun 1;217(6):e20200652. doi: 10.1084/jem.20200652. PMID 32302401
- [Result] Narasaraju T, Tang BM, Herrmann M, Muller S, Chow VTK, Radic M. Neutrophilia and NETopathy as Key Pathologic Drivers of Progressive Lung Impairment in Patients With COVID-19. Front Pharmacol. 2020 Jun 5;11:870. doi: 10.3389/fphar.2020.00870. eCollection 2020. PMID 32581816
- [Result] de Wilde AH, Raj VS, Oudshoorn D, Bestebroer TM, van Nieuwkoop S, Limpens RWAL, Posthuma CC, van der Meer Y, Barcena M, Haagmans BL, Snijder EJ, van den Hoogen BG. MERS-coronavirus replication induces severe in vitro cytopathology and is strongly inhibited by cyclosporin A or interferon-alpha treatment. J Gen Virol. 2013 Aug;94(Pt 8):1749-1760. doi: 10.1099/vir.0.052910-0. Epub 2013 Apr 25. PMID 23620378
- [Result] Softic L, Brillet R, Berry F, Ahnou N, Nevers Q, Morin-Dewaele M, Hamadat S, Bruscella P, Fourati S, Pawlotsky JM, Ahmed-Belkacem A. Inhibition of SARS-CoV-2 Infection by the Cyclophilin Inhibitor Alisporivir (Debio 025). Antimicrob Agents Chemother. 2020 Jun 23;64(7):e00876-20. doi: 10.1128/AAC.00876-20. Print 2020 Jun 23. PMID 32376613